CLINICAL TRIAL: NCT00566176
Title: Thoracoscopically-Assisted Epicardial Bilateral Pulmonary Vein Isolations Using the AtriCure Bipolar System and Exclusion of the Left Atrial Appendage for the Treatment of Atrial Fibrillation
Brief Title: Sole-Therapy Treatment of Atrial Fibrillation
Acronym: RESTORE SR II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2005-1
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; AF; AFIB; racing heart; pulmonary vein isolation; pvi; mini maze; maze
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia

INTERVENTIONS:
Device: Surgical Ablation using the AtriCure Bipolar System — Surgical Ablation using the AtriCure Bipolar System

SUMMARY:
RESTORE SR II is a feasibility study on the minimally invasive use of the AtriCure Bipolar System for PV Isolation on a beating heart for the treatment of all types of atrial fibrillation in a sole therapy operation (not concomitant to another cardiac operation).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient between 18 and 80 years of age
2. Patient with symptomatic AF and failure or intolerance of one or more Class I or Class III AADs and:

   * Who describes 3 or more symptomatic AF episodes during the 6 month period prior to enrollment, with at least 1 electrocardiographically documented episode of AF in the 4 months prior to enrollment or,
   * Who has documented AF within the 6 months proceeding enrollment that did not terminate spontaneously (including patients in continuous AF) or,
   * Who is unwilling or unable to take anticoagulants, with 3 or more symptomatic episodes during the 6 month period prior to enrollment with at least 1 electrocardiographically documented episode of AF in the 4 months prior to enrollment.
3. Left Atrial Size < 6 cm (determined by echocardiography performed within 60 days of enrollment), unless the LV dysfunction is thought to result (at least in part) from AF
4. Left Ventricular Ejection Fraction ≥ 30% (determined by echocardiography performed within 60 days of enrollment)
5. Patient is willing and able to provide written informed consent.
6. Patient has a life expectancy of at least 2 years.
7. Patient is willing and able to attend the scheduled follow-up visits.
8. Weight < 325 lbs

Exclusion Criteria:

1. Prior cardiac catheter ablation for the treatment of arrhythmia within 4 months
2. Prior cardiac surgery
3. Patients requiring any open heart procedure (e.g. CABG, valve replacement or repair, atrial septal defect repair, etc.)
4. Class IV NYHA heart failure symptoms, unless these symptoms are considered to be due to uncontrolled AF
5. Cerebrovascular accident within previous 6 months
6. Known carotid artery stenosis greater than 80%
7. Evidence of significant active infection
8. Patient unable to undergo TEE
9. Pregnant woman
10. Requires anti-arrhythmic drug therapy for the treatment of ventricular arrhythmia
11. Presence of thrombus in the left atrium
12. Patient has co-morbid condition that in the opinion of the investigator poses undue risk of general anesthesia or port access cardiac surgery
13. Patient is enrolled in another investigational study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the feasibility of performing this operation by demonstrating the ability to consistently isolate the right and left PVs using this minimally invasive approach. | Perioperatively
The primary safety endpoint will be determined by assessing the rate of serious adverse events. | Discharge/30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Warren Jackman, MD, Principal Investigator — University of Oklamhoma Cardiac Arrythmia Research Institute; James Edgerton, MD, Principal Investigator — Medical City Hospital/Cardio Pulmonary Research Science and Technology Institute
Locations (5):
- United States (5):
  - University Community Hospital/Dr. Kiran C. Patel Research Institute, Tampa, Florida
  - University of Cincinnati, Cincinnati, Ohio
  - University of Oklahoma Cardiac Arrythmia Research Institute, Oklahoma City, Oklahoma
  - Sacred Heart Medical Center Endovascular Research, Eugene, Oregon
  - Medical City Hospital/Cardio Pulmonary Research Science and Technology Institute, Dallas, Texas